CLINICAL TRIAL: NCT07328672
Title: Investigation of the Effects of Pain Neuroscience Education and Basic Body Awareness Therapy on Pain, Autonomic Nervous System Responses, and Pelvic Floor Muscle Activity in Women With Chronic Pelvic Pain
Brief Title: Pain Neuroscience Education and Basic Body Awareness Therapy in Women With Chronic Pelvic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sena Öndeş (Other)
Collaborators: Istinye University (Other)
Responsible Party: Sponsor-Investigator, Sena Öndeş, Lecturer, Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DrThesis
Record Dates: First submitted 2025-11-25; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pelvic Pain Syndrome; Female
Keywords: Body Awareness; Basic Body Awareness Therapy; Pelvic Floor Muscle Activity; Autonomic Nervous System; Physiotherapy; Rehabilitation; Chronic Pelvic Pain; Pelvic Floor Muscles; Pain Neuroscience Education
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Neuroscience Education + Standard Physiotherapy and Rehabilitation (Experimental): Participants receive the standard physiotherapy and rehabilitation program in addition to structured Pain Neuroscience Education sessions.
  Interventions: Behavioral: Standard Physiotherapy and Rehabilitation; Behavioral: Pain Neuroscience Education
- Basic Body Awareness Therapy + Standard Physiotherapy Group (Experimental): Participants receive the standard physiotherapy and rehabilitation program in addition to Basic Body Awareness Therapy sessions focusing on posture, movement and breathing.
  Interventions: Behavioral: Standard Physiotherapy and Rehabilitation; Behavioral: Basic Body Awareness Therapy
- Standard Physiotherapy and Rehabilitation Group (Active Comparator): Participants receive standard pelvic physiotherapy and rehabilitation interventions, including relaxation training, myofascial release, stretching, breathing, and aerobic exercises.
  Interventions: Behavioral: Standard Physiotherapy and Rehabilitation

INTERVENTIONS:
Behavioral: Standard Physiotherapy and Rehabilitation — The interventions will be conducted over 8 weeks, with sessions held twice per week.
  The Standard Physiotherapy and Rehabilitation program includes pelvic floor muscle relaxation, myofascial release, stretching, breathing and relaxation exercises, and aerobic training.
Behavioral: Pain Neuroscience Education — The Pain Neuroscience Education (PNE) group will receive the same physiotherapy program plus weekly educational sessions focused on pain neurophysiology, central sensitization, and cognitive reframing strategies, delivered by a physiotherapist trained in Pain Neuroscience Education.
  Arms: Pain Neuroscience Education + Standard Physiotherapy and Rehabilitation
Behavioral: Basic Body Awareness Therapy — The Basic Body Awareness Therapy (BBAT) group will receive the same physiotherapy program plus weekly body awareness sessions emphasizing postural alignment, movement control and breathing. Exercises will be practiced in supine, sitting, and standing positions to enhance body-mind awareness.
  All interventions will be supervised by an experienced pelvic floor physiotherapist at Istinye University.
  Arms: Basic Body Awareness Therapy + Standard Physiotherapy Group

SUMMARY:
This randomized controlled trial aims to investigate the effects of Pain Neuroscience Education and Basic Body Awareness Therapy, when added to standard physiotherapy and rehabilitation, on pain, autonomic nervous system responses, and pelvic floor muscle activity in women with chronic pelvic pain. A total of 45 women diagnosed with chronic pelvic pain will be randomly allocated into three groups: (1) standard physiotherapy and rehabilitation, (2) standard physiotherapy plus Pain Neuroscience Education, and (3) standard physiotherapy plus Basic Body Awareness Therapy. The study will assess pain intensity (algometry, NRS, SF-MPQ), pain catastrophizing, autonomic responses (electrodermal activity), pelvic floor muscle activation (EMG), and related psychological, cognitive, and body awareness parameters. Secondary outcomes will include sexual function, quality of life, and patient satisfaction. The aim is to compare two awareness-based interventions-one primarily mind-to-body (Pain Neuroscience Education) and the other body-to-mind (Basic Body Awareness Therapy)-to determine their relative and complementary effects on pain perception and physiological regulation in women with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Women with any type of chronic pelvic pain, including pelvic floor muscle dysfunction, endometriosis, vulvodynia, genito-pelvic pain/penetration disorder, or bladder pain syndrome, with pain persisting for six months or longer.

Exclusion Criteria:

* Presence of pelvic infections, inflammatory conditions, or pelvic malignancy.
* Pregnancy.
* History of urogynecological surgery within the last six months.
* Presence of advanced pelvic organ prolapse.
* Patients currently receiving chemotherapy or radiotherapy.
* Patients whose primary complaint is not chronic pelvic pain.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women diagnosed with chronic pelvic pain will be eligible to participate in this study. Male participants are excluded because the interventions and outcome measures are specifically designed for female pelvic floor function and related disorders.
Enrollment: 45 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold and Pain Tolerance | Baseline and up to 8 weeks
  Pressure pain threshold and tolerance will be assessed using a Baseline® manual algometer. Standardized measurement points will be located in the abdominal and pelvic regions (15 points in total). Pressure will be applied perpendicularly at a rate of 1 kg/s until the participant reports the first pain sensation and maximum tolerable pain. The mean of two measurements per site will be used for analysis. Distal control points (C5-C6 zygapophyseal level, second metacarpal, and tibialis anterior muscle) will be included to evaluate widespread pressure sensitivity as an indicator of central sensitization.
Pain Intensity and Characteristics (Short Form McGill Pain Questionnaire) | Baseline and up to 8 weeks
  Pain intensity and characteristics will be assessed using the Short Form McGill Pain Questionnaire (SF-MPQ). The SF-MPQ evaluates both sensory (11 items) and affective (4 items) dimensions of pain through 15 descriptors rated on a 4-point scale (0 = none to 3 = severe). It also includes a Visual Analog Scale (VAS) and a 6-point Likert scale assessing overall pain intensity (0 = no pain to 5 = unbearable pain). Total scores will be calculated for sensory, affective, and overall dimensions.
Pain Catastrophizing (Pain Catastrophizing Scale) | Baseline and up to 8 weeks
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), a 13-item self-report questionnaire developed by Sullivan et al. to measure negative cognitive and emotional responses to pain. Each item is rated on a 5-point Likert scale (0 = not at all, 4 = all the time), with total scores ranging from 0 to 52. Higher scores indicate greater levels of catastrophizing. The PCS includes three subscales: rumination, magnification, and helplessness.
Autonomic Nervous System Responses - Tonic Skin Conductance Level (SCL) | Baseline and up to 8 weeks
  Resting tonic skin conductance level will be recorded using the Shimmer3 GSR+ device with electrodes placed on the hypothenar region. Higher SCL indicates increased sympathetic arousal.
Autonomic Nervous System Responses- Phasic Skin Conductance Response (SCR) Amplitude | Baseline and up to 8 weeks
  Phasic SCR amplitude will be recorded during painful pressure stimuli applied at the Pfannenstiel incision point. This parameter reflects rapid sympathetic responses to pain.
Autonomic Nervous System Responses- Skin Conductance Response Frequency | Baseline and up to 8 weeks
  The total number of phasic responses during the stimulus period will be counted to quantify response frequency.
Autonomic Nervous System Responses- Skin Conductance Response Latency | Baseline and up to 8 weeks
  Latency from stimulus onset to the first SCR will be measured to assess autonomic response timing.
Resting Pelvic Floor Muscle Activity (Resting sEMG) (Surface Electromyography) | Baseline and up to 8 weeks
  Resting pelvic floor muscle activity will be recorded using surface electromyography (NeuroTrac® MyoPlus PRO). Electrodes will be placed bilaterally in the perianal region. Mean resting µV value across trials will be used for analysis.
Minimum Pelvic Floor Muscle Activation (Minimum sEMG) (Surface Electromyography) | Baseline and up to 8 weeks
  Minimum muscle activation during contraction attempts will be recorded in µV. The lowest activation value across the contraction-relaxation cycles will be used.
Maximum Voluntary Contraction of Pelvic Floor Muscles (MVC) (Surface Electromyography) | Baseline and up to 8 weeks
  MVC will be assessed during five maximal pelvic floor contractions. Values will be expressed as percent activation relative to baseline.
Pelvic Floor Muscle Relaxation Time (Surface Electromyography) | Baseline and up to 8 weeks
  Relaxation time will be measured as the time required for sEMG amplitude to return from peak activation to baseline following a contraction.

SECONDARY OUTCOMES:
Pain-Related Beliefs (Pain Beliefs Questionnaire) | Baseline and up to 8 weeks
  Pain-related cognitive beliefs will be assessed using the Pain Beliefs Questionnaire (PBQ), which evaluates individuals' beliefs about the causes, meaning, and controllability of pain. The PBQ consists of two subscales: organic beliefs (the idea that pain indicates tissue damage) and psychological beliefs (the idea that pain is influenced by emotional and mental processes). Each item is rated on a 6-point Likert scale (1 = never, 6 = always), with higher scores indicating stronger beliefs in each domain. The questionnaire will be used to assess changes in pain-related cognitions and cognitive restructuring following the interventions.
Pelvic Floor Symptoms (Global Pelvic Floor Bother Questionnaire) | Baseline and up to 8 weeks
  Pelvic floor dysfunction-related symptoms will be assessed using the Global Pelvic Floor Bother Questionnaire (PFBQ). This questionnaire evaluates the severity of pelvic floor symptoms and their impact on daily life, including stress urinary incontinence, urinary frequency, urgency, urge incontinence, voiding difficulty, pelvic organ prolapse, obstructive defecation, fecal incontinence, and dyspareunia. Each symptom is answered as "Yes/No," and if "Yes," participants rate the bother level from 1 (not at all) to 5 (a lot). The total score ranges from 0 to 45, with higher scores indicating greater symptom severity or bother.
Female Sexual Function (Female Sexual Function Index) | Baseline and up to 8 weeks
  Female sexual function will be assessed using the Female Sexual Function Index (FSFI), a validated, multidimensional questionnaire developed by Rosen et al. It consists of 19 items rated on a 5-point Likert scale and evaluates six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Total scores range from 2.0 to 36.0, with higher scores indicating better sexual function. A cutoff score of 26.55 differentiates between normal and dysfunctional sexual function.
Depression, Anxiety, and Stress Levels (Depression Anxiety Stress Scale-21) | Baseline and up to 8 weeks
  Depression, anxiety, and stress levels will be assessed using the Depression Anxiety Stress Scale-21 (DASS-21), a reliable 21-item self-report questionnaire developed by Lovibond & Lovibond and validated in Turkish by Yılmaz et al. (2017). The scale includes three subscales-depression, anxiety, and stress-each with seven items rated on a 4-point Likert scale (0 = did not apply to me at all to 3 = applied to me very much). Higher scores indicate greater emotional distress. Severity for each subscale is categorized as normal, mild, moderate, severe, or extremely severe.
Interoceptive Awareness (Multidimensional Assessment of Interoceptive Awareness II) | Baseline and up to 8 weeks
  Interoceptive awareness will be evaluated using the Multidimensional Assessment of Interoceptive Awareness II (MAIA-II), developed by Mehling et al. (2018) and validated in Turkish by Özpınar et al. (2021). The MAIA-II consists of 37 items rated on a 6-point Likert scale (0 = never to 5 = always) and measures eight dimensions of interoceptive awareness, including noticing, attention regulation, emotional awareness, self-regulation, and body trust. Higher scores indicate greater interoceptive awareness. Negatively worded items (items 5-12 and 15) are reverse-scored before subscale means are calculated.
Quality of Life (WHOQOL-BREF) | Baseline and up to 8 weeks
  Quality of life will be evaluated using the World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF) and the Pelvic Pain Impact Questionnaire (PIQ). The WHOQOL-BREF, validated in Turkish by Eser et al. (1999), consists of 27 items rated on a 5-point Likert scale and assesses four domains: physical, psychological, social, and environmental. Higher scores indicate better quality of life.
Quality of Life (Pelvic Pain Impact Questionnaire) | Baseline and up to 8 weeks
  The PIQ, developed by Chalmers et al. (2017) and validated in Turkish by Kurt et al. (2023), is an 8-item Likert-type scale assessing the multidimensional impact of chronic pelvic pain on energy, mood, sleep, gastrointestinal function, sitting tolerance, daily activities, physical activity, and clothing. Two additional open-ended questions address sexual activity and tampon use but are not included in the total score. Higher scores reflect greater impact of pain on daily life.
Patient Satisfaction (Numeric Rating Scale) | After 8 weeks of intervention
  Patient satisfaction with the treatment will be assessed using a Numeric Rating Scale (NRS). Participants will be asked to rate their overall satisfaction with the treatment on a scale from 0 to 10, where 0 indicates "not satisfied at all" and 10 indicates "completely satisfied." Higher scores reflect greater satisfaction. This subjective self-assessment will be conducted at the end of the 8-week intervention period.